CLINICAL TRIAL: NCT01757275
Title: A Multi-center, Randomised, Double-blind, Parallel-group Phase III Study to Assess High Dose Esomeprazole Na i.v. Treatment (Bolus Infusion of 80 mg Followed by a Continuous Infusion of 8 mg Per Hour Administered for 72 Hours) for Prevention of Rebleeding
Brief Title: High Dose Esomeprazole Na for Prevention of Rebleeding After Successful Endoscopic Therapy of a Bleeding Peptic Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D961DC00007
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Bleeding Peptic Ulcer
Keywords: peptic ulcer bleeding; prevention of rebleeding; successful endoscopic haemostatic therapy
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Esomeprazole; Cimetidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Esomeprazole (Experimental)
  Interventions: Drug: Esomeprazole Na; Drug: Esomeprazole Mg
- Cimetidine (Active Comparator)
  Interventions: Drug: Cimetidine

INTERVENTIONS:
Drug: Esomeprazole Na — Given as 80mg bolus infusion during 30 min and then 8mg/h constant infusion during 71.5 hous
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Cimetidine — Given as 200mg bolus infusion during 30 min and then 60mg/h constant infusion during 71.5 hours
  Arms: Cimetidine
Drug: Esomeprazole Mg — 40 mg tablet once daily for 27 days
  Other Names: Nexium
  Arms: Esomeprazole

SUMMARY:
To describe the rate of clinically significant rebleeding during 72 hours continuous i.v. infusion of high dose esomeprazole Na in patients in China with primary successful endoscopic haemostatic therapy of a bleeding peptic ulcer, with cimetidine i.v. in

DETAILED DESCRIPTION:
A multi-center, randomised, double-blind, parallel-group phase III study to assess high dose esomeprazole Na i.v. treatment (bolus infusion of 80 mg followed by a continuous infusion of 8 mg per hour administered for 72 hours) for prevention of rebleeding

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Female or male aged =18 years and =70 years.
* Acute upper gastrointestinal bleeding (haematemesis, melaena or haematochezia) or such signs within the last 24 hours as judged by the investigator.
* One endoscopically confirmed bleeding gastric or duodenal peptic ulcer, at least 5 mm in diameter, classified as Forrest Ia, Ib, IIa, or IIb. Photo documentation of the source of bleeding should be provided.
* Successful haemostasis (which is considered to have been established if bleeding has stopped and, if applicable, formerly bleeding vessels are flattened or cavitated) achieved by endoscopic treatment and confirmed by site staff.

Exclusion Criteria:

* Endoscopic suspicion of gastric malignancy or juxta pyloric stenosis as judged by the investigator.
* Sign of multi PUB or concomitant other gastro bleeding from esophageal varices, reflux esophagitis, gastritis, Mallory Weiss rifts, ulcus simplex, Dieulafoy's lesion, colon, small bowel, or ulcer distal to the stom in Billroth-resected patients.
* Need for treatment during the first 7 days of the study with NSAIDs, Cyclooxygenase-2 (COX-2) inhibitors, acetyl salicylic acid (ASA) (including low dose) or clopidogrel.
* Planned treatment with: warfarin (including other vitamin K antagonists), cisapride, phenytoin, atazanavir, nelfinavir, digoxin, methotrexate, clopidogrel, tacrolimus, theophylline, lidocaine, nifedipine.
* Chemotherapy or radiation therapies within 2 weeks prior to randomisation or planned during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca Molndal, Sweden
Locations (12):
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Ha'er Bing
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an

REFERENCES:
- [Derived] Bai Y, Chen DF, Wang RQ, Chen YX, Shi RH, Tian DA, Chen H, Eklund S, Li ZS; Chinese Peptic Ulcer Bleeding Research Group. Intravenous Esomeprazole for Prevention of Peptic Ulcer Rebleeding: A Randomized Trial in Chinese Patients. Adv Ther. 2015 Nov;32(11):1160-76. doi: 10.1007/s12325-015-0265-6. Epub 2015 Nov 18. PMID 26581750
- See also: China_PUB_Study_D961DC00007_Clinical_Study_Protocol_GEL_Redacted_(approved) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=690&filename=China_PUB_Study_D961DC00007_Clinical_Study_Protocol_GEL_Redacted_(approved).pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 239 patients were enrolled from 19 centres in China. The first patient entered the study on 26 February 2013 and the last patient completed the study on 30 December 2014.
  Of the 239 patients enrolled into the study, 222 (92.9%) patients were randomised to treatment.
Pre-assignment Details: 17 patients were not assigned to treatment, 15 patients did not fulfil the eligibility criteria, 1 was due to patient decision, and 1 patient due to "other" (not enough experimental drug).
Groups:
- Esomeprazole: Esomeprazole iv 80 mg bolus infusion for 30 min followed by Esomeprazole iv 8 mg/hour for 71.5 hours and esomeprazole oral 40 mg once daily for 27 days
- Cimetidine: Cimetidine iv 200 mg bolus infusion for 30 min followed by Cimetidine iv 60 mg/hour for 71.5 hours and esomeprazole oral 40 mg once daily for 27 days
Period: Overall Study
Arm/Group | Esomeprazole | Cimetidine
Started | 111 | 111
Completed | 102 | 98
Not Completed | 9 | 13
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Not treated | 3 | 4

BASELINE CHARACTERISTICS:
Population: Among 222 randomised patients, 215 patients received iv treatment: 108 patients in the esomeprazole treatment group and 107 patients in the cimetidine treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Cimetidine | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 42.4 (12.79) | 41.8 (12.96) | 42.1 (12.85)
Age, Customized [Number; unit: participants]
  <=65 years | 104 | 103 | 207
  >65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 83 | 83 | 166
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Chinese | 108 | 107 | 215
Number of patients with one bleeding ulcer [Number; unit: participants] | 108 | 107 | 215
Forrest class [Number; unit: participants] — Forrest classification of PUB (Forrest et al 1974): Ia = arterial bleeding; Ib = oozing bleeding; IIa = non-bleeding visible vessel; IIb = adherent clot.
  participants
    Ia | 5 | 4 | 9
    Ib | 58 | 64 | 122
    IIa | 33 | 24 | 57
    IIb | 12 | 15 | 27
Bleeding ulcer size [Mean (Standard Deviation); unit: mm] | 8.2 (4.8) | 8.1 (3.6) | 8.1 (4.3)
Ulcer location [Number; unit: participants]
  Stomach | 17 | 8 | 25
  Duodenum | 84 | 89 | 173
  Stomach and Duodenum | 7 | 10 | 17
Number of patients with ulcers of different sizes [Number; unit: participants]
  <=2 cm | 105 | 106 | 211
  >2 cm | 3 | 1 | 4
Number of patients with single and multiple ulcers [Number; unit: participants]
  Single | 89 | 89 | 178
  Multiple | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinically Significant Rebleeding Within 72 Hours
Description: Diagnostic criteria for clinically significant rebleeding based on either A, B or C:
  A) Endoscopy - initiated by clinical signs of bleeding defined as one of B1 or B2 or B3 and endoscopic verification, ie one of A1 or A2.
  A1: Blood in stomach (this criteria cannot be used during the first 6 hours after primary endoscopic haemostasis). A2: A verified active bleeding from a peptic ulcer (Forrest Ia, Ib).
  B) A true clinically based definition, at least two of B1 and/or B2 and/or B3. B1: Vomiting of fresh blood or fresh blood in a gastric tube or haematochezia or melaena after a normal stool. B2: Decrease in Hb >20g/L (or Hct >6%) during 24 hours or an increase in Hb <10g/L (or Hct <3%) despite ≥2 units of blood has been transfused during 24hours. B3: Unstable circulation systolic blood pressure ≤ 90 mmHg or pulse ≥110/min (after have had a stable circulation).
  C) Haematemesis. Vomiting significant amounts (>200 ml) of fresh blood as estimated by the investigator.
Time Frame: 72 hours
Population: Full analysis set (FAS). All randomised patients, who started the randomised iv treatment (bolus dose), were included in the FAS.
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No rebleeding | 107 | 101
  Rebleeding | 1 | 6

2. Secondary Outcome: Rate of Clinically Significant Rebleeding During 7 Days
Description: as for outcome 1
Time Frame: 7 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No rebleeding | 105 | 101
  Rebleeding | 3 | 6

3. Secondary Outcome: Rate of Clinically Significant Rebleeding During 30 Days
Description: as for outcome 1
Time Frame: 30 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No rebleeding | 105 | 101
  Rebleeding | 3 | 6

4. Secondary Outcome: Number of Patients With Endoscopic Re-treatment Within 72 Hours
Time Frame: 72 hours
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No re-treatment | 108 | 106
  Re-treatment | 0 | 1

5. Secondary Outcome: Number of Patients With Endoscopic Re-treatment Within 30 Days
Time Frame: 30 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No re-treatment | 106 | 106
  Re-treatment | 2 | 1

6. Secondary Outcome: Number of Patients With Surgery Due to Rebleeding Within 72 Hours
Time Frame: within 72 hours
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No surgery | 108 | 107
  Surgery | 0 | 0

7. Secondary Outcome: Number of Patients With Surgery Due to Rebleeding Within 30 Days
Time Frame: within 30 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
participants
  No surgery | 108 | 106
  Surgery | 0 | 1

8. Secondary Outcome: Number of Blood Units Transfused Within 72 Hours
Time Frame: within 72 hours
Population: FAS
Measure: Number; unit: blood units
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
blood units | 14 | 21

9. Secondary Outcome: Number of Blood Units Transfused Within 30 Days
Time Frame: within 30 days
Population: FAS
Measure: Number; unit: blood units
Arm/Group | Esomeprazole | Cimetidine
Number analyzed (Participants) | 108 | 107
blood units | 18 | 21

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of the first administration of IP until the end of study, up to 35 days. SAEs will be collected from signed inform consent until the end of the study, up to 36 days.
Arm/Group | Esomeprazole | Cimetidine
Serious Adverse Events (participants affected / at risk) | 5/110 | 5/105
Other Adverse Events (participants affected / at risk) | 22/110 | 20/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole (N=110) | Cimetidine (N=105)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=110) | Cimetidine (N=105)
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Persecutory delusion (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Blood fibrinogen decreased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Neutrophil percentage increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1

LIMITATIONS AND CAVEATS:
No hypothesis testing was performed in this study and, as such, no formal statistical comparisons were made. Two patients who were initially randomised to receive cimetidine treatment actually received esomeprazole treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No